CLINICAL TRIAL: NCT02769871
Title: Effect of Showing Stroke Neuroimaging to Patients in Setting of Smoking Cessation Education on Smoking Cessation Rates in Patients With New Stroke.
Brief Title: NICE: NeuroImaging in Cessation Education
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of team members.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1606017908
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2019-06

CONDITIONS: Stroke; Smoking Cessation
MeSH Terms: conditions — Stroke; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Standardized smoking cessation counseling (Active Comparator): Standardized smoking cessation counseling will be provided at the participant's initial interview. Participants will be provided pamphlets from the National Stroke Association and the American Heart Association regarding risk factor reduction. Packets will include general information on risks associated with smoking along with the benefits of cessation, and methods to quit. Pamphlets will include Life's Simple 7 (American Heart Association, 2014) and Be Smoke Free: Facts about Smoking and Stroke Risk (National Stroke Association, 2009). Counseling will be scripted and standardized to ensure similar language with all participants.
  Interventions: Behavioral: standardized smoking cessation counseling
- Neuroimages of stroke (Experimental): Participants in the intervention group will undergo standardized smoking cessation counseling (as offered to the active comparator group) and will also be shown computer images of head CT or brain MRI (DWI/FLAIR series) of their strokes. Basic orientation to neuroimaging (laterality, positioning, parts of the brain) will be provided first, and then the image of the stroke itself will be reviewed. Participants will be provided with a paper copy of the slice demonstrating the largest volume of stroke to keep. In comparison, participants will also be shown images of a normal healthy, and images of a patient with recurrent strokes due to smoking. Participants will be told that smoking cessation would help to prevent additional stroke, but that it would not repair the damage already done, as visualized on the neuroimaging.
  Interventions: Behavioral: Neuroimages of stroke

INTERVENTIONS:
Behavioral: Neuroimages of stroke — Participants in the intervention group will be shown computer images of head CT or brain MRI (DWI/FLAIR series) of their strokes. Basic orientation to neuroimaging (laterality, positioning, parts of the brain) will be provided first, and then the image of the stroke itself will be reviewed. Participants will be provided with a paper copy of the slice demonstrating the largest volume of stroke to keep. In comparison, patients will also be shown images of a normal healthy, and images of a patient with recurrent strokes due to smoking. Patients will be told that smoking cessation would help to prevent additional stroke, but that it would not repair the damage already done, as visualized on the neuroimaging.
  Arms: Neuroimages of stroke
Behavioral: standardized smoking cessation counseling — Standardized smoking cessation counseling will be provided at their initial interview. They will be provided pamphlets from the National Stroke Association and the American Heart Association regarding risk factor reduction. Packets will include general information on risks associated with smoking along with the benefits of cessation, and methods to quit. Pamphlets will include Life's Simple 7 (American Heart Association, 2014) and Be Smoke Free: Facts about Smoking and Stroke Risk (National Stroke Association, 2009). Counseling will be scripted and standardized to ensure similar language with all participants.
  Arms: Standardized smoking cessation counseling

SUMMARY:
The investigators aim to examine the effect on smoking cessation rate by showing stroke patients who are active smokers images of their strokes.

DETAILED DESCRIPTION:
The investigators hypothesize that showing actual images of a patient's stroke to the participant on either brain CT or MRI will be a similarly easy to understand quantification of damage done to the participant's body. Given the link between smoking and stroke risk, the investigators believe that providing this imaging in addition to standard smoking cessation education may improve rates of smoking cessation after stroke. If this proves true, addition of a patient's neuroimaging to standard post-stroke smoking cessation education would be an easy method to improve smoking cessation rates in stroke patients, at minimal cost.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Active smoker, as defined: at least 100 cigarettes in their entire life, must have smoked cigarette at least once in 4 days prior to onset of stroke
* Primary ischemic or hemorrhagic stroke identified on neuroimaging (MRI DWI/ADC or CT of brain)
* Onset of stroke symptoms within 30 days to time of recruitment
* Capacity to comprehend counseling data: Each participant will be given a cognitive screening test to assess the ability to comprehend and accurately answer the medical history questionnaire (MMSE). If the participant fails this test (score < 23), they will be excluded.
* Patients discharged home or short term rehab with expectation of returning home within the study period

Exclusion Criteria:

* Patients whose stroke deficits clinically prevent them from reasonably being physically able to continue to smoke, such as bilateral upper extremity paresis, tracheostomy, GCS ≥9
* Patients with sensory aphasia that impairs comprehension
* Subarachnoid hemorrhage
* Transient ischemic attack
* Other cause of cerebral ischemia or hemorrhage not defined as primary ischemic or hemorrhagic stroke (i.e. hemorrhagic metastases)
* Patients whose stroke symptoms started >30 days from time of enrollment
* Patients discharged to acute rehab, long term acute care hospital or hospice who are unlikely to have access to cigarettes
* Patients unable to complete cognitive screening test for whom an appropriate proxy does not exist
* Patients who do not speak fluent English (given that the study largely revolves around oral education on smoking cessation, clear communication between participant and coordinator must be possible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
cessation of smoking measured by self-report collected during follow-up phone interviews. | 30 day follow-up visit
  30 day and 90 day post-stroke phone interviews will be by a blinded APRN. During these interviews, patients will be asked their smoking status. If they are still smoking, they will be asked how much they are still smoking,
cessation of smoking measured by self-report collected during follow-up phone interviews. | 90 day follow-up visit
  30 day and 90 day post-stroke phone interviews will be by a blinded APRN. During these interviews, patients will be asked their smoking status. If they are still smoking, they will be asked how much they are still smoking,

SECONDARY OUTCOMES:
number of cigarettes smoked per day measured by self-report collected during follow-up phone interviews. | 30 day follow-up visit
  30 day and 90 day post-stroke phone interviews will be by a blinded APRN. During these interviews, patients will be asked their smoking status. If they are still smoking, they will be asked how much they are still smoking,
number of cigarettes smoked per day measured by self-report collected during follow-up phone interviews. | 90 day follow-up visit
  30 day and 90 day post-stroke phone interviews will be by a blinded APRN. During these interviews, patients will be asked their smoking status. If they are still smoking, they will be asked how much they are still smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Hardik Amin, MD, Principal Investigator — Yale University

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082